CLINICAL TRIAL: NCT00212251
Title: Promoting Postpartum Weight Loss in Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00012546; R01DK064986 (NIH); DK64986; Duke IRB #4399
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: obesity; postpartum period; exercise; diet; motivation
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Diet, Fat-Restricted

ARMS (1):
- Lifestyle counseling (Experimental): 10 ActiveMoms classes, 8 Moms Time Out nutrition classes, 6 coaching calls, supportive materials
  Interventions: Behavioral: moderate exercise and healthy, low-fat diet

INTERVENTIONS:
Behavioral: moderate exercise and healthy, low-fat diet

SUMMARY:
The purpose of this study is to evaluate, in a five-year randomized controlled trial, the efficacy of an intervention (AMP - ACTIVE MOTHERS POSTPARTUM) to increase physical activity and promote a healthy diet (decreased calorie and fat intake) for weight loss among postpartum women who were overweight or obese prior to pregnancy. The hypothesis is that the proportion of women losing at least 10% of BMI from baseline to 12 months post-intervention will be significantly greater in the AMP intervention arm than in the minimal care arm.

DETAILED DESCRIPTION:
Retention of weight gained in pregnancy contributes to the development of overweight and obesity in middle age, now at epidemic proportions in America. While interventions to reduce weight retention specifically targeting the postpartum period have been few, interventions that promote modest weight loss starting in early postpartum are safe and could be efficacious, particularly for women who were overweight prior to pregnancy. Moreover, postpartum-related changes in cognitive factors (risk perceptions), behavioral factors (physical activity, diet), self concept (self-esteem) and social role (work, food preparation, child care) may make this time a "teachable moment" that could be capitalized upon by formal interventions. Interventions could leverage natural weight changes to encourage adoption of a healthy diet and increase physical activity, which together could accelerate and/or increase natural weight loss in postpartum. Whether the postpartum period is a teachable moment for weight loss interventions can be investigated empirically.

ELIGIBILITY:
Inclusion Criteria:

* pre-pregnancy BMI>24
* over 18
* delivered baby in past 6 weeks
* English speaking
* driving distance to Duke University Medical Center

Exclusion Criteria:

* Hemodynamically significant heart disease
* Restrictive lung disease
* Severe anemia
* Unevaluated maternal cardiac arrythmia
* Chronic bronchitis
* Poorly controlled Type 1 diabetes
* Poorly controlled hypertension
* Orthopedic limitations
* Poorly controlled seizure disorder
* Poorly controlled hyperthyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-08; Study Completion 2008-04

PRIMARY OUTCOMES:
BMI change from baseline to 12 months post-intervention (24 months postpartum) will be assessed via self-report and validated by in-person weight measurement. The proportion of women who lose 10% of baseline BMI

SECONDARY OUTCOMES:
Change in BMI from pre-pregnancy to 12 months post-intervention; proportion below their pre-pregnancy weight at 1, 6 and 12 months post-intervention; and BMI change from baseline to 1 a

CONTACTS AND LOCATIONS:
Overall Officials: Truls Ostbye, MD, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Ostbye T, Krause KM, Brouwer RJ, Lovelady CA, Morey MC, Bastian LA, Peterson BL, Swamy GK, Chowdhary J, McBride CM. Active Mothers Postpartum (AMP): rationale, design, and baseline characteristics. J Womens Health (Larchmt). 2008 Dec;17(10):1567-75. doi: 10.1089/jwh.2007.0674. PMID 19049350
- [Result] Ostbye T, Krause KM, Lovelady CA, Morey MC, Bastian LA, Peterson BL, Swamy GK, Brouwer RJ, McBride CM. Active Mothers Postpartum: a randomized controlled weight-loss intervention trial. Am J Prev Med. 2009 Sep;37(3):173-80. doi: 10.1016/j.amepre.2009.05.016. PMID 19595557
- [Derived] Durham HA, Morey MC, Lovelady CA, Namenek Brouwer RJ, Krause KM, Ostbye T. Postpartum physical activity in overweight and obese women. J Phys Act Health. 2011 Sep;8(7):988-93. doi: 10.1123/jpah.8.7.988. PMID 21885890
- [Derived] Durham HA, Lovelady CA, Brouwer RJ, Krause KM, Ostbye T. Comparison of dietary intake of overweight postpartum mothers practicing breastfeeding or formula feeding. J Am Diet Assoc. 2011 Jan;111(1):67-74. doi: 10.1016/j.jada.2010.10.001. PMID 21185967
- [Derived] Krause KM, Lovelady CA, Ostbye T. Predictors of breastfeeding in overweight and obese women: data from Active Mothers Postpartum (AMP). Matern Child Health J. 2011 Apr;15(3):367-75. doi: 10.1007/s10995-010-0667-7. PMID 20821042